CLINICAL TRIAL: NCT01208623
Title: A Large Series of Clinical and Imaging Investigation to Patients With Chronic Lower Limb Edema With Unclear Etiology
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Wing P. Chan, Wan Fang Hospital Department of Radiology
Other Study IDs: NSC99-2314-B-038-024-; 99040 (Other: WF IRB)
Record Dates: First submitted 2010-09-20; First posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Lower Limb Edema With Unclear Etiology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 2D: 2D digital venography images alone
- 3D: 3D rotational venography
- Combine: combined MDCT angiography/venography

SUMMARY:
Patients with chronic lower limb edema commonly suffered from extremities edema, pain, varicosities, venous stasis changes, and deep venous thrombosis. A common challenge for primary care physicians is to determine the cause and find an effective treatment for leg edema of unclear etiology. The aims of this project are to determine the cause of patients with chronic lower limb edema with conventional digital venography, the clinical value of role of 3D rotational venography or combined multidetector (MD)CT angiography and iliac venography using direct iliac venography for contrast administration via bilateral femoral catheterization (MDCT angiography/venography) with volume-rendering images supplementary to 2D digital venography in evaluation of patients with chronic lower limb edema.

This project is designed as retrospective cross-sectional study. Between April 2008 and Dec 2009, a total of approximately 300 patients with chronic lower limb edema who had had bilateral iliac digital venography and surgery at our institution will be reviewed. All patients underwent surgery by one senior vascular surgeon for lower limb conditions within one month after the venographic examination. Patients who had incomplete clinical and surgical records or incomplete images will be excluded. The surgical findings of the presence, anatomical location, and size of the venous narrowing will assessed and described. Stenosis was defined as luminal narrowing of 50% or more compared to the prestenotic or poststenotic lumen.With use of surgical findings as a the standard, the investigators calculated and compared the diagnostic accuracies, sensitivities, specificities, positive predict values and negative predict values of 2D digital venography images alone, 3D rotational venography, and combined MDCT angiography/venography with volume-rendering images supplementary to 2D digital venography.

With this large series study, the investigators believe that the cause of chronic lower leg edema in our patients' population will be clarified. The value of additional 3D rotational venography, and combination MDCT angiography/venography with volume-rendering images will lead to higher diagnostic performance and may provide a helpful tool for planning surgical and endovascular treatment, which has not been reported before.

DETAILED DESCRIPTION:
Patients with chronic lower limb edema commonly suffered from extremities edema, pain, varicosities, venous stasis changes, and deep venous thrombosis. A common challenge for primary care physicians is to determine the cause and find an effective treatment for leg edema of unclear etiology. The aims of this project are to determine the cause of patients with chronic lower limb edema with conventional digital venography, the clinical value of role of 3D rotational venography or combined multidetector (MD)CT angiography and iliac venography using direct iliac venography for contrast administration via bilateral femoral catheterization (MDCT angiography/venography) with volume-rendering images supplementary to 2D digital venography in evaluation of patients with chronic lower limb edema.

This project is designed as retrospective cross-sectional study. Between April 2008 and Dec 2009, a total of approximately 300 patients with chronic lower limb edema who had had bilateral iliac digital venography and surgery at our institution will be reviewed. All patients underwent surgery by one senior vascular surgeon for lower limb conditions within one month after the venographic examination. Patients who had incomplete clinical and surgical records or incomplete images will be excluded. The surgical findings of the presence, anatomical location, and size of the venous narrowing will assessed and described. Stenosis was defined as luminal narrowing of 50% or more compared to the prestenotic or poststenotic lumen.With use of surgical findings as a the standard, we calculated and compared the diagnostic accuracies, sensitivities, specificities, positive predict values and negative predict values of 2D digital venography images alone, 3D rotational venography, and combined MDCT angiography/venography with volume-rendering images supplementary to 2D digital venography.

With this large series study, we believe that the cause of chronic lower leg edema in our patients' population will be clarified. The value of additional 3D rotational venography, and combination MDCT angiography/venography with volume-rendering images will lead to higher diagnostic performance and may provide a helpful tool for planning surgical and endovascular treatment, which has not been reported before.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had complete clinical and surgical records or incomplete images.

Exclusion Criteria:

* Patients who had incomplete clinical and surgical records or incomplete images.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between April 2008 and Dec 2009, a total of approximately 300 patients with chronic lower limb edema who had had bilateral iliac digital venography and surgery at our institution will be reviewed. All patients underwent surgery by one senior vascular surgeon for lower limb conditions within one month after the venographic examination.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wing P. Chan, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan